CLINICAL TRIAL: NCT01286103
Title: An Open-Label, Multiple-Dose Study to Assess the Steady-State Pharmacokinetics, Pharmacodynamics and Safety of Once-Daily Versus Twice-Daily Dosing With Canagliflozin in Healthy Subjects
Brief Title: A Pharmacokinetic and Pharmacodynamic Study of Once-Daily and Twice-Daily Dosing With Canagliflozin in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Director, Clinical Pharmacology Leader, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017824; 28431754DIA1032
Record Dates: First submitted 2011-01-13; First posted 2011-01-31 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: Canagliflozin; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Canagliflozin

ARMS (2):
- 001 (Experimental): Canagliflozin 300 mg once daily and 150 mg twice daily Treatment A (one 300-mg tablet once daily for 5 days) followed 10 days later by Treatment B (one 50-mg and one 100-mg tablet twice daily for 5 days) or Treatment B followed by Treatment A.
  Interventions: Drug: Canagliflozin 300 mg once daily and 150 mg twice daily
- 002 (Experimental): Canagliflozin 100 mg once daily and 50 mg twice daily Treatment C (one 100-mg tablet once daily for 5 days) followed 10 days later by Treatment D (one 50-mg tablet twice daily for 5 days) or Treatment D followed by Treatment C.
  Interventions: Drug: Canagliflozin 100 mg once daily and 50 mg twice daily

INTERVENTIONS:
Drug: Canagliflozin 300 mg once daily and 150 mg twice daily — Treatment A (one 300-mg tablet once daily for 5 days) followed 10 days later by Treatment B (one 50-mg and one 100-mg tablet twice daily for 5 days) or Treatment B followed by Treatment A.
  Arms: 001
Drug: Canagliflozin 100 mg once daily and 50 mg twice daily — Treatment C (one 100-mg tablet once daily for 5 days) followed 10 days later by Treatment D (one 50-mg tablet twice daily for 5 days) or Treatment D followed by Treatment C.
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the effects of canagliflozin on glucose levels in the blood and urine when taken at 2 dose levels as a once-daily or twice-daily dosing regimen in healthy adult volunteers

DETAILED DESCRIPTION:
This is an open-label (volunteers will know the names of treatments they are assigned), single-center study of canagliflozin (JNJ-28431754) in healthy adult volunteers. Canagliflozin (a Sodium-Glucose Cotransporter 2 inhibitor) is currently under development to lower blood sugar levels in patients with type 2 diabetes mellitus (T2DM). Patients in Cohort 1 will be randomized to receive Treatment A (one 300-mg tablet orally, by mouth [PO] once daily for 5 days) followed 10 days later by Treatment B (one 50-mg and one 100-mg tablet PO twice daily for 5 days) or Treatment B followed by Treatment A. Patients in Cohort 2 will be randomized to receive Treatment C (one 100-mg tablet PO once daily for 5 days) followed 10 days later by Treatment D (one 50-mg tablet PO twice daily for 5 days) or Treatment D followed by Treatment C.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index (BMI, a measure of a person's weight in relation to height) between 18 and 30 kg/m2, inclusive, and a body weight of not less than 50 kg

Exclusion Criteria:

* History of or current clinically significant medical illness as determined by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose
* Known allergy to canagliflozin or any of the excipients of the formulation of canagliflozin

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-01; Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin | Up to Day 5 after the last treatment
Plasma concentrations of glucose | Up to Day 5 after the last treatment
Urinary glucose excretion (UGE) | Up to Day 5 after the last treatment
Renal threshold of glucose (RTG) | Up to Day 5 after the last treatment

SECONDARY OUTCOMES:
The number and type of adverse events reported | Up to 10 days after last dose (last dose is given on Day 8)
Changes in hematology laboratory parameters | Up to 10 days after last dose (last dose is given on Day 8)
Changes in chemistry laboratory parameters | Up to 10 days after last dose (last dose is given on Day 8)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Devineni D, Polidori D, Curtin CR, Murphy J, Wang SS, Stieltjes H, Wajs E. Pharmacokinetics and pharmacodynamics of once- and twice-daily multiple-doses of canagliflozin, a selective inhibitor of sodium glucose co-transporter 2, in healthy participants. Int J Clin Pharmacol Ther. 2015 Jun;53(6):438-46. doi: 10.5414/CP202324. PMID 25907176